CLINICAL TRIAL: NCT01005940
Title: Health Outcomes of Treatment of Obstructive Sleep Apnea With Dental Devices
Brief Title: Dental Device for Treatment of Sleep Apnea
Acronym: OSA-MAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulysses Magalang MD (Other)
Responsible Party: Sponsor-Investigator, Ulysses Magalang MD, Professor-Clinical, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2009H0131
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2021-07

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep Apnea Syndromes; Insulin Resistance; Mandibular advancement device
MeSH Terms: conditions — Sleep Apnea Syndromes; Insulin Resistance | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mandibular advancement device (Experimental): Subject is evaluated when receiving intervention with mandibular advancement device.
  Interventions: Device: Mandibular advancement device
- No mandibular advancement device (No Intervention): Subject is evaluated when not receiving treatment with mandibular advancement device.

INTERVENTIONS:
Device: Mandibular advancement device — Mandibular advancement device made to subject specific specifications
  Arms: Mandibular advancement device

SUMMARY:
This study is being done to see if treatment of obstructive sleep apnea (OSA) with a mandibular advancement device (MAD) shows an increase in the quality of life. Many patients prefer to call them mandibular advancers, jaw advancers, jaw advancement splints, jaw advancement devices, anti-snoring mouthpieces, or oral appliances for the treatment of snoring and mild to moderate obstructive sleep apnea. The investigators will also see how helpful the mandibular advancement device is on insulin resistance.

DETAILED DESCRIPTION:
Patients with obstructive sleep apnea (OSA) will be included in this prospective controlled trial. OSA patients who are unable to tolerate CPAP or refuse CPAP(Continuous positive airway pressure) (and who are deemed appropriate by their attending physician for dental device treatment of OSA will be randomized to a control group (no MAD treatment) or to active MAD therapy.

Epidemiologic studies suggest that OSA is associated with insulin resistance independent of other known risk factors such as obesity. The cyclic intermittent hypoxia in OSA is the primary stimulus that leads to insulin resistance, a primary risk factor for the development of type 2 diabetes. There is an association between the level of hypoxic stress in OSA and insulin resistance.

The overall hypothesis to be tested is that treatment of OSA with MAD will improve insulin sensitivity, increase levels of HMW (High-molecular- weight) adiponectin, and improve psychological adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Apnea-hypopnea index (AHI) of at least 20 events/hr based on overnight polysomnography
* > 18 years of age
* Unable to tolerate or refuse CPAP treatment

Exclusion Criteria:

* Known diabetes mellitus
* Body mass index (BMI) > 45 kg/m2
* Uncontrolled hypertension
* Known congestive heart failure
* Use of illicit drugs
* Excessive alcohol consumption, defined as:

  * More than 3 glasses of wine a day
  * More than 3 beers a day
  * More than 60 mL of hard liquor a day
* Room air oxyhemoglobin saturation < 90%
* Use of home oxygen
* Use of corticosteroids
* Unable to give voluntary consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Treatment of OSA with mandibular advancement device results in improvements in insulin sensitivity | 16 weeks

SECONDARY OUTCOMES:
Treatment of OSA with mandibular advancement device increases the levels of high-molecular-weight adiponectin in the circulation | 16 weeks
Treatment of OSA with mandibular advancement device improves psychological adjustment. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses Magalang, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No